CLINICAL TRIAL: NCT04459884
Title: Multicenter Observational Study on Practice of Ventilation in Brain Injured Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: VENTIBRAIN
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Mechanical Ventilation; Acute Brain Injury
MeSH Terms: conditions — Brain Injuries | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: mechanical ventilation — mechanical ventilation > 48h

SUMMARY:
Rationale Several experimental and clinical studies have shown how brain injury can cause secondary lung injury. Lung injury could be due either to mechanical ventilation- often necessary in brain injured patients- or to inflammatory response that follows primary acute brain injury. The concept of 'Protective lung ventilation' has shown to reduce morbidity and mortality of intensive care unit (ICU) patients with acute respiratory distress syndrome (ARDS) but seems also to have a beneficial effect on patients with healthy lungs and in the perioperative settings. However, these recommendations often come into conflict with the management of patients affected by acute brain injury, in which permissive hypercapnia and increased intrathoracic pressure as consequence of protective ventilation strategies can be dangerous.

Study design This is an international multi-center prospective observational study.

Study population This study will include all consecutive brain injured patients (traumatic brain injury (TBI) or cerebrovascular) intubated and ventilated in ICU and observed for a 7-day period.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness Seen the observational design of the study, there is no patient burden. Collection of data from ICU and hospital charts and/or (electronic) medical records systems is of no risk to patients.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE Mechanical ventilation (MV) is a frequently applied and often a life-saving strategy in neurocritically ill patients. Paradoxically, ventilation itself has the potential to cause further pulmonary and cerebral damage and can increase mortality and morbidity [1].

The so-called 'protective lung ventilation' strategies include the use of low tidal volume (TV), positive end expiratory pressure (PEEP), and eventually recruitment maneuvers (RMs), and are aimed to prevent lung damage and to reduce morbidity and mortality in patients with acute respiratory distress syndrome (ARDS) [2]. In particular, low tidal volume seems to have the greater importance [3-5], and guidelines strongly recommend its use in critically ill patients with ARDS [6].

Results from one multicenter randomized controlled trial suggest that also ICU patients without ARDS could benefit from 'protective lung ventilation strategies [7]. A recent meta-analysis showed a higher incidence of pulmonary complications and even increased mortality in patients who received 'conventional ventilation' with traditionally sized or higher tidal volumes compared to patients undergoing protective strategies [8].

Present ventilation guidelines for patients with acute brain injury The fourth edition of the Guidelines for the Management of Severe Traumatic Brain Injury [10] suggests maintaining normocapnia in this subset of patients and aiming for peripheral saturation of oxygen higher than 90% to guarantee an adequate cerebral perfusion and avoid secondary brain damages due to hypoxia or inappropriate cerebral vasodilatation [10]. However, BTF guidelines do not provide any advice on ventilator settings or targets. There is still uncertainty regarding the use of protective ventilation in neurologically ill patients. Brain injured patients have been traditionally excluded from the major trials regarding mechanical ventilation and the use of lung protective ventilator strategies because low tidal volumes, high PEEP and RMs can increase carbon dioxide levels (CO2) and increase intrathoracic pressure, thus having detrimental effects on intracranial pressure (ICP) and cerebral perfusion pressure (CPP).

METHODS

Objectives

This observational study aims to determine the ventilation practice of consecutive intubated and ventilated neuro-ICU patients in the first week from admission in intensive care units.

Hypotheses

* In patients with acute brain injury, protective ventilation strategies are not often applied; in particular, tidal volumes are higher than those used in patients with no brain injury. The adoption of protective ventilation in this group of patients might result in a beneficial effect on outcome.
* Ventilation practice, in particular tidal volume size, varies among patients with acute brain injury and among different centers and different countries.
* In patients with acute brain injury outcomes can be dependent on ventilator setting.

Study design

International multicenter prospective observational study of consecutive ventilated neuro-ICU patients in the first week since admission to ICU.

Study population

We will collect data of consecutive patients with acute brain injury intubated and ventilated, admitted to the intensive care unit (ICU).

Sample size calculation

The primary endpoint of the study is the exploration of the ventilator settings in clinical practice in braininjured patients. The hypotheses of the study are exploratory; hence a sample size calculation has not been conducted. This international prospective observational study aims to recruit>3000 patients in coma after acute brain damage admitted to >200 Intensive Care Units (ICUs). Recruitment will last 12 weeks at each center, aiming to enroll about 20 patients/center. To avoid any overrepresentation of some centers we ceil the data collection to 30 patients/center. This number of enrolled patients and ICUs reflects an adequate sample size to capture a range of variation in practice between ICUs. We aim to include also low-middle income countries, in order to have a representation of the variability worldwide.

Follow-up/Outcomes

Enrolled patients will be followed until ICU-discharge or death (whatever comes first), for collection of patient demographics (on day of admission), and ventilation characteristics (from start of ventilation till stop of ventilation). At 6 months, data on length of hospital stay and outcome (Extended Glasgow Coma Scale) will be collected.

Outcomes will be assessed as:

* 6-months mortality and neurological outcome (as for extended Glasgow Outcome Scale, eGOS)
* Hospital length of stay (in days), in hospital mortality.
* Mortality, duration of mechanical ventilation (in days), ventilator free days (days) at ICU discharge.

Study procedures

Patients in participating centers are screened on a daily basis. ICU-patients under mechanical ventilation and with diagnosis of acute brain injury will be included. Demographic data on screened patients regardless of meeting enrollment criteria will be recorded (registry).

The inclusion period will be flexible for participating centers and determined at a later stage together with the study-coordinator.

Times points of data collection

* Demographic data and baseline data, including severity scores (e.g. APACHE II- scores and SAPS III) will be collected from clinical files on the day of start of mechanical ventilation.
* Ventilation settings, gas exchange variables and vital parameters will be collected once daily in the morning till the day when ventilation is stopped or till day 7, whichever comes first.
* Chest radiography data from available chest X-rays (i.e., no extra chest X-rays are obtained) in the first week.
* Lung echography data are collected from clinical files in the first week.
* Predefined complications are recorded from medical chart (Appendix 1)
* At ICU discharge: mortality, duration of mechanical ventilation (in days), ventilator free days (days).
* At 6-months: mortality and neurological outcome (as for extended Glasgow Outcome Scale, eGOS), length of stay (in days), in hospital mortality.

Inclusion During a 3 months period, all admitted patients will be screened daily by a local investigator.

STATISTICAL ANALYSIS

Patient characteristics will be compared and described by appropriate statistics. Student's t-test or Mann-Whitney U-tests will be used to compare continuous variables and chi-squared tests will be used for categorical variables. Data will be expressed as means (SD), medians (interquartile range) and proportions as appropriate. Comparisons between and within groups will be performed using one-way ANOVA and post-hoc analyses for continuous variables.

Plan of analysis The primary analysis will concern the determination of (variation of) the ventilator settings in neurologically critically ill patients. Univariate analysis will be performed to identify potential factors associated with outcomes including, but not limited to, GOS, mortality, duration of ventilation, or hospital LOS. A multivariate logistic regression model will be used to identify independent risk factors. A stepwise approach will be used to enter new terms into the model, with a limit of p < 0.2 to enter the terms. Time to event variables will be analyzed using Cox regression and visualized by Kaplan-Meier. Statistical analyses will be conducted using R. A p value of less than 0.05 was considered statistically significant.

ETHICAL CONSIDERATIONS Ethical standards The PI and Steering Committee will ensure that this study is conducted in full conformity with the Declaration of Helsinki and Good Clinical Practices.

Ethics committee Each NC/PI will notify the relevant ethics committee, in compliance with the local legislation and rules. The national coordinators will facilitate this process. The approval of the protocol (if required by local authorities) must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the SC before the changes are implemented to the study.

Lack of capacity and Delayed Consent Informed consent will be obtained from patients with no lack of capacity. For patients not be able to provide informed consent at the time of recruitment, the responsible clinical/research staff will act as Consulter and consent eligible patients after discussion with the next- of-kin.If the patient has a Power of Attorney or a Legal tutor or an, he/she will act as Consultee and will be asked to consent/decline participation to the study on legal behalf of the patient.

If patients have Advance Decision Plan including participation in research studies the Plan will be respected and recruitment pursued/abandoned accordingly. At follow-up, patients who have regained capacity will be asked to provide Informed Consent and will be given the possibility to:

* Provide Informed Consent for the acute data and follow-up.
* Deny research participation and request destruction of acute data collected.

Expected impact of the study The investigators expect to obtain data of >3000 patients admitted to ICU. These data will allow a detailed description of patient's characteristics, management strategies resource use and correlation with clinical outcomes. In particular, the study will provide insights in relation to clinical management, monitoring and treatment, practice variation in neurointensive care units around the world, differences in the ventilator management of brain injured patients and their potential association with outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the ICU with a diagnosis of

  * traumatic brain injury or
  * cerebrovascular diseases (intracranial hemorrhage, subarachnoid hemorrhage, ischemic stroke)
* Patients requiring intubation and mechanical ventilation in the ICU
* Expected ventilation for more than 48 hours

Exclusion Criteria:

* Age < 18 years
* Pregnant patients
* Patients not intubated or not mechanically ventilated or receiving only non-invasive ventilation (i.e., the patient never received invasive ventilation during the present admission)
* Patients under invasive mechanical ventilation before the 7-day period of inclusion
* Expected ventilation or death< 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will collect data of consecutive patients with acute brain injury intubated and ventilated, admitted to the intensive care unit (ICU).
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Description of different ventilatory strategies applied to acutely brain injured patients admitted to the ICUs | 12 months
  We will compare the different ventilatory approaches to intubated and mechanically ventilated neurocritically ill patients admitted to worldwide ICUs.

SECONDARY OUTCOMES:
Correlation between ventilatory targets and neurological outcome at ICU discharge and after 6 months from admission | 12 months
  We explore the correlation of ventilator settings and targets with outcome in the whole population (neurological outcome Glasgow Outcome Scale Extended)
Description of different ventolatory approaches to nuerocritically-ill patients | 12 months
  The differences in ventilator settings among different countries will be described
Description of mechanical ventilation-associated complication | 12 months
  We will describe the incidence of pulmonary complications (including pneumonia, ARDS, neurogenic pulmonary edema) in the whole cohort of patients
Correlation between ventilatory targets and neurological secondary injury | 12 months
  We will describe the ventilator settings applied when intracranial pressure is raised (>20 mmHg) and we will describe the need for adjustments related to intracranial hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Robba, MD, Principal Investigator — University of Milano Bicocca
Locations (1):
- ASST-Monza, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: No
Data collection will be web-based. Participating centres will collect data via an electronic Case-Report Form (REDCAP cloud); data will be automatically pseudoanonymized with a numeric alpha code; the list of correspondence between the patient's code and its identity will be stored in a safe place and access to this data will be granted only to study PI and study staff delegated by the PI and listed in the delegation log. The data resides at the University of Milano-Bicocca. The study will be conducted in accordance with the Helsinki Declaration and in accordance with the rules of Good Clinical Practice (D.M. Healthcare of 15/07/1997 and s.m.i.) as well as with the applicable regulatory provisions.
  The patient's personal data will be processed in accordance with the European Personal Data Protection Regulation (GDPR), Di.Lgs. 196/2003 and subsequent changes and additions, and any other Italian law applicable to the protection of personal data.

REFERENCES:
- [Result] Slutsky AS. Lung injury caused by mechanical ventilation. Chest. 1999 Jul;116(1 Suppl):9S-15S. doi: 10.1378/chest.116.suppl_1.9s-a. No abstract available. PMID 10424561
- [Result] Putensen C, Theuerkauf N, Zinserling J, Wrigge H, Pelosi P. Meta-analysis: ventilation strategies and outcomes of the acute respiratory distress syndrome and acute lung injury. Ann Intern Med. 2009 Oct 20;151(8):566-76. doi: 10.7326/0003-4819-151-8-200910200-00011. PMID 19841457
- [Result] Esteban A, Ferguson ND, Meade MO, Frutos-Vivar F, Apezteguia C, Brochard L, Raymondos K, Nin N, Hurtado J, Tomicic V, Gonzalez M, Elizalde J, Nightingale P, Abroug F, Pelosi P, Arabi Y, Moreno R, Jibaja M, D'Empaire G, Sandi F, Matamis D, Montanez AM, Anzueto A; VENTILA Group. Evolution of mechanical ventilation in response to clinical research. Am J Respir Crit Care Med. 2008 Jan 15;177(2):170-7. doi: 10.1164/rccm.200706-893OC. Epub 2007 Oct 25. PMID 17962636
- [Result] Matthay MA, Ware LB, Zimmerman GA. The acute respiratory distress syndrome. J Clin Invest. 2012 Aug;122(8):2731-40. doi: 10.1172/JCI60331. Epub 2012 Aug 1. PMID 22850883
- [Result] Needham DM, Colantuoni E, Mendez-Tellez PA, Dinglas VD, Sevransky JE, Dennison Himmelfarb CR, Desai SV, Shanholtz C, Brower RG, Pronovost PJ. Lung protective mechanical ventilation and two year survival in patients with acute lung injury: prospective cohort study. BMJ. 2012 Apr 5;344:e2124. doi: 10.1136/bmj.e2124. PMID 22491953
- [Result] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Result] Determann RM, Royakkers A, Wolthuis EK, Vlaar AP, Choi G, Paulus F, Hofstra JJ, de Graaff MJ, Korevaar JC, Schultz MJ. Ventilation with lower tidal volumes as compared with conventional tidal volumes for patients without acute lung injury: a preventive randomized controlled trial. Crit Care. 2010;14(1):R1. doi: 10.1186/cc8230. Epub 2010 Jan 7. PMID 20055989
- [Result] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Result] Neto AS, Barbas CSV, Simonis FD, Artigas-Raventos A, Canet J, Determann RM, Anstey J, Hedenstierna G, Hemmes SNT, Hermans G, Hiesmayr M, Hollmann MW, Jaber S, Martin-Loeches I, Mills GH, Pearse RM, Putensen C, Schmid W, Severgnini P, Smith R, Treschan TA, Tschernko EM, Melo MFV, Wrigge H, de Abreu MG, Pelosi P, Schultz MJ; PRoVENT; PROVE Network investigators. Epidemiological characteristics, practice of ventilation, and clinical outcome in patients at risk of acute respiratory distress syndrome in intensive care units from 16 countries (PRoVENT): an international, multicentre, prospective study. Lancet Respir Med. 2016 Nov;4(11):882-893. doi: 10.1016/S2213-2600(16)30305-8. Epub 2016 Oct 4. PMID 27717861
- [Result] Carney N, Totten AM, O'Reilly C, Ullman JS, Hawryluk GW, Bell MJ, Bratton SL, Chesnut R, Harris OA, Kissoon N, Rubiano AM, Shutter L, Tasker RC, Vavilala MS, Wilberger J, Wright DW, Ghajar J. Guidelines for the Management of Severe Traumatic Brain Injury, Fourth Edition. Neurosurgery. 2017 Jan 1;80(1):6-15. doi: 10.1227/NEU.0000000000001432. PMID 27654000
- [Result] Picetti E, Pelosi P, Taccone FS, Citerio G, Mancebo J, Robba C; on the behalf of the ESICM NIC/ARF sections. VENTILatOry strategies in patients with severe traumatic brain injury: the VENTILO Survey of the European Society of Intensive Care Medicine (ESICM). Crit Care. 2020 Apr 17;24(1):158. doi: 10.1186/s13054-020-02875-w. PMID 32303255
- [Result] Gajic O, Dabbagh O, Park PK, Adesanya A, Chang SY, Hou P, Anderson H 3rd, Hoth JJ, Mikkelsen ME, Gentile NT, Gong MN, Talmor D, Bajwa E, Watkins TR, Festic E, Yilmaz M, Iscimen R, Kaufman DA, Esper AM, Sadikot R, Douglas I, Sevransky J, Malinchoc M; U.S. Critical Illness and Injury Trials Group: Lung Injury Prevention Study Investigators (USCIITG-LIPS). Early identification of patients at risk of acute lung injury: evaluation of lung injury prediction score in a multicenter cohort study. Am J Respir Crit Care Med. 2011 Feb 15;183(4):462-70. doi: 10.1164/rccm.201004-0549OC. Epub 2010 Aug 27. PMID 20802164
- [Result] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Derived] Robba C, Citerio G, Taccone FS, Galimberti S, Rebora P, Vargiolu A, Pelosi P; VENTIBRAIN Enlarged Steering committee members; VENTIBRAIN. Multicentre observational study on practice of ventilation in brain injured patients: the VENTIBRAIN study protocol. BMJ Open. 2021 Aug 11;11(8):e047100. doi: 10.1136/bmjopen-2020-047100. PMID 34380722